CLINICAL TRIAL: NCT01073631
Title: Post Marketing Surveillance Study To Observe The Safety And Efficacy Of Vfend® Tablet
Brief Title: Non-Interventional Post Marketing Surveillance Study To Observe The Safety And Efficacy Of Vfend® Tablet In Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1501068
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2010-09-13 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-05

CONDITIONS: Serious Fungal Infections
Keywords: voriconazole; Korea; invasive fungal infection
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients who are indicated for use of voriconazole tablet.
  Interventions: Drug: voriconazole tablet

INTERVENTIONS:
Drug: voriconazole tablet — 200 mg PO bid (orally, twice a day)
  Other Names: Vfend

SUMMARY:
This is a non-interventional study of voriconazole tablet in Korea which is mandated by the Korean government agency.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated for voriconazole table according to the drug package insert.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are indicated for voriconazole tablet according to the drug package insert.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501068&StudyName=Non-Interventional%20Post%20Marketing%20Surveillance%20Study%20To%20Evaluate%20The%20Safety%20And%20Efficacy%20Of%20Vfend%AE%20Tablet%20In%20Korea%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 543 participants enrolled in this study. Of these, 230 participants were treated with the Vfend tablet formulation only, and 313 participants were treated with Vfend tablet and Vfend intravenous (IV) formulations sequentially or vice versa. These 313 participants are also included in Study A1501067 (NCT01073618).
Groups:
- Vfend: Vfend (voriconazole) tablets (recommended dose: 200mg orally every 12hours) or sequential Vfend tablet and IV Vfend (recommended dose: 6mg/kg IV infusion every 12hours for first 24hours [loading dose], 3 to 4mg/kg IV infusion every 12hours [maintenance dose]) treatment (or vice versa) for use as indicated according to approved local product document and adjusted according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Vfend
Started | 543
Completed | 374
Not Completed | 169
Not completed — Death | 82
Not completed — Adverse Event | 24
Not completed — Other | 63

BASELINE CHARACTERISTICS:
Arm/Group | Vfend
Number analyzed (Participants) | 543
Age, Customized [Number; unit: Participants]
  <18 years | 74
  Between 18 and 44 years | 157
  Between 45 and 64 years | 207
  >=65 years | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 332

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Categorical Clinical Response: Cure, Improvement, Failure, or Unevaluable
Description: Clinical response defined as: Cure=resolution of all baseline signs and symptoms of fungal infection(s); Improvement=lessening of baseline signs and symptoms or absence of one or more, but not all baseline findings; Failure=no improvement or deterioration of baseline condition; Unevaluable=incomplete therapy (efficacy could not be evaluated or discontinuation was not followed up).
Time Frame: Baseline (Day 1) up to 2.1 Years
Population: Safety population: participants received at least 1 dose of study drug for approved indication (= Intent to treat [ITT] population plus all unevaluable participants); ITT=participants received study drug for the approved indication and had been evaluated for related paramenters at least once.
Measure: Number; unit: Percentage of participants
Arm/Group | Vfend
Number analyzed (Participants) | 543
Percentage of participants
  Cure | 36.83
  Improvement | 26.52
  Failure | 16.94
  Unevaluable | 19.71
Statistical Analysis 1: Comparison: Vfend; Efficacy Rate (treatment effective) = Percentage of evaluable participants with clinical response of cure or improvement; Test type: Superiority or Other; Normal approximation to binomial; Efficacy rate (percent) = 78.90, 95% CI 2-sided [75.07 to 82.73] — Confidence Interval (CI) by normal approximation to binomial

2. Secondary Outcome: Percentage of Participants With Cultivated Strain Mycological Response: Eradication, Persistence, Superinfection, or Not Evaluable
Description: In case cultivation performed, cultivated strain before and after Vfend administration recorded, and the improvement of mycological outcomes after administration evaluated. Mycological response defined as: Eradication=absence of signs and symptoms of fungal infection; Persistence=(no eradication) presence of fungal infection; Superinfection=existence of different strains from strains separated prior to study treatment; Not evaluable=a follow-up mycological cultivation not performed.
Time Frame: Baseline (Day 1) up to 2.1 Years
Population: ITT; N=number of participants evaluated for mycological response.
Measure: Number; unit: Percentage of participants
Arm/Group | Vfend
Number analyzed (Participants) | 88
Percentage of participants
  Eradication | 71.59
  Persistence | 23.86
  Superinfection | 2.27
  Not evaluable | 2.27

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from the time of the first dose of study treatment up to 28 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Vfend
Serious Adverse Events (participants affected / at risk) | 119/543
Other Adverse Events (participants affected / at risk) | 154/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vfend (N=543)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Neutropenic colitis (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 3
Multi-organ failure (General disorders) | 6
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Acute graft versus host disease in intestine (Immune system disorders) | 2
Acute graft versus host disease in skin (Immune system disorders) | 2
Anal abscess (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 21
Pneumonia staphylococcal (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 15
Septic shock (Infections and infestations) | 18
Cytomegalovirus test positive (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 2
Grand mal convulsion (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Haemorrhage (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Euthyroid sick syndrome (Endocrine disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Central nervous system infection (Infections and infestations) | 1
Citrobacter sepsis (Infections and infestations) | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1
Acoustic stimulation tests (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vfend (N=543)
Anaemia (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 7
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Atrial fibrillation (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Otorrhoea (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Eye disorder (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Keratoconjunctivitis sicca (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 3
Visual impairment (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oesophagitis (Gastrointestinal disorders) | 1
Perianal erythema (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Chest discomfort (General disorders) | 1
Feeling abnormal (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 18
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Acute graft versus host disease in intestine (Immune system disorders) | 2
Graft versus host disease (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 1
Anal abscess (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 5
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 6
Infection (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase (Investigations) | 1
Blood bilirubin increased (Investigations) | 2
Blood creatine increased (Investigations) | 2
Blood creatinine increased (Investigations) | 4
Blood test (Investigations) | 1
Blood urea increased (Investigations) | 4
Haemoglobin decreased (Investigations) | 2
Immunosuppressant drug level increased (Investigations) | 1
Liver function test abnormal (Investigations) | 9
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Transaminases increased (Investigations) | 5
White blood cell count decreased (Investigations) | 3
White blood cell count increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Major depression (Psychiatric disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 1
Angina pectoris (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.